CLINICAL TRIAL: NCT06804590
Title: A Randomized, Double-blind, Parallel-group, Phase III Study to Compare the Clinical Efficacy, Safety, and Immunogenicity of Denosumab Injection 9MW0311 With Prolia® in Postmenopausal Women With Osteoporosis
Brief Title: A Study on Efficacy, Safety and Immunogenicity of 9MW0311 in Postmenopausal Women With Osteoporosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW0311-2024-CP302
Record Dates: First submitted 2024-12-09; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Postmenopausal Women Osteoporosis
Keywords: Denosumab; efficacy; MW031; postmenopausal women; safety
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW0311 (Experimental): 9MW0311 Denosumab injection(60 mg)
  Interventions: Drug: 9MW0311
- Prolia® (Active Comparator): Prolia® Denosumab injection(60 mg)
  Interventions: Drug: Prolia®

INTERVENTIONS:
Drug: 9MW0311 — 9MW0311 Denosumab injection(60 mg) was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Arms: 9MW0311
Drug: Prolia® — Prolia® Denosumab injection(60 mg) was administered subcutaneously once every 6 months for a maximum of 2 consecutive doses throughout the trial.
  Arms: Prolia®

SUMMARY:
This study is a multicenter, randomized, double-blinded, parallel-group Phase III clinical study to compare the clinical efficacy, safety, and immunogenicity of 9MW0311 and Prolia® in Chinese postmenopausal women with osteoporosis at high risk for fracture.

DETAILED DESCRIPTION:
278 patients are randomized 1:1 to receive 9MW0311 and Prolia® every 6 months for 12 months. The primary efficacy endpoint is the percentage change from baseline in BMD at the lumbar spine(LS) in month 12.

ELIGIBILITY:
Inclusion Criteria:

* Women who can walk freely (≥50 and ≤80 years);
* As measured by DXA, the absolute value of BMD at lumbar spine, femoral neck or total hip was -4.0<T value ≤-2.5;
* Subjects must have at least one of the following other risk factors: 1) history of previous fragility fractures; 2) Either or both parents have a history of hip fragility fracture; 3) Increased bone turnover rate during screening; 4) Low body weight; 5) Old age(≥70); 6) Currently smoking.
* The duration of spontaneous amenorrhea was >2 years or >2 years after bilateral oophorectomy. If the status of bilateral oophorectomy is unknown or if the ovaries are preserved after hysterectomy, follicle stimulating hormone (FSH) levels >40mIU/mL may be used to confirm the status of postoperative menopause.

Exclusion Criteria:

* Bone/metabolic disease
* Hyperparathyroidism or hypoparathyroidism
* Thyroid condition: Hyperthyroidism or hypothyroidism
* Rheumatoid arthritis
* Malignant tumors
* Malabsorption syndrome
* Liver cirrhosis, active hepatitis B or hepatitis C, and unstable liver disease; serum aspartate aminotransferase and alanine aminotransferase ≥ 2.0 times the upper limit of normal (ULN); alkaline phosphatase or total bilirubin ≥ 1.5 ULN;
* Renal disease - severe impairment of kidney function
* Clinically significant cardiovascular and cerebrovascular diseases (such as myocardial infarction, unstable angina or stroke, NYHA class III or IV heart failure in the 12 months prior to screening) and hematopoietic system disease judged by the investigator;
* Hypercalcemia or hypocalcemia ;
* vitamin D deficiency (25-hydroxyvitamin D, 25OHD <20 ng/mL);
* Oral or dental diseases: previous or current evidence of mandibular osteomyelitis or osteonecrosis; Acute dental or mandibular disease requiring oral surgery; Planning invasive dental surgery; Failure to recover from dental or oral surgery;
* Use of intravenous bisphosphonates within the previous 2 years;
* oral bisphosphonates (used for at least 2 years, or used for less than 2 years but more than 3 months, with the last use occurring <1 year before the screening);
* Use of any of the following drugs within 6 weeks prior to screening that may affect bone metabolism:

  1. parathyroid hormone (PTH) or PTH derivatives, such as teriparatide;
  2. anabolic hormones or testosterone;
  3. glucocorticoids (equivalent dose more than 5mg/ day of prednisone and continuous use for more than 10 days);
  4. Selective estrogen receptor modulators (SERMs), such as raloxifene;
  5. Menopausal hormone therapy (such as estrogen, estrogen + progesterone, tibolone);
  6. Active vitamin D and its analogues (cumulative use of more than 30 days);
  7. Other bone-active drugs include antiepileptic drugs (except benzodiazepines) and heparin;
  8. Long-term systemic use of ketoconazole, adrenocorticotropin (ACTH), aluminum, lithium, protease inhibitors, methotrexate, gonadotropin releasing hormone agonists;
  9. Chinese patent medicines for osteoporosis related treatment are clearly described in the instructions, such as Xianling Gubao capsule (tablet), Gushukang capsule (granule), Jintiange capsule and Qianggu capsule."
* History of more than two vertebral fractures.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 278 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in lumbar spine(LS)-BMD at Week 53 （Month 12) | Baseline and 12 months
  Percent Change From Baseline in LS-BMD at Week 53 （Month 12)

SECONDARY OUTCOMES:
Percent Change From Baseline in LS-BMD at Week 27 （Month 6) | Baseline and Month 6
  Percent Change From Baseline in LS-BMD at Week 27 （Month 6)
Percent change in BMD at the total hip, femoral neck from Baseline up to week 27 (Month 6) and Week 53 (Month 12 ) | Baseline, Month6 and Month 53
  Percent change in BMD at the total hip, femoral neck from Baseline up to week 27 (Month 6) and Week 53 (Month 12 )
Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) and Serum type I procollagen N-terminal propeptide (s-PINP) from Baseline up to 12 months | Baseline, Month1, Month3, Month6, Month9 and Month 12
  Percent Change in Serum Carboxy-terminal Cross-linking Telopeptide of Type I Collagen (s-CTX) and Serum type I procollagen N-terminal propeptide (s-PINP) from Baseline up to 12 months
Proportion of subjects with new fragility fractures (e.g., vertebrae, hip, non-vertebrae) | From baseline to Month12
  Proportion of subjects with new fragility fractures (e.g., vertebrae, hip, non-vertebrae)
Number of participants with AE, SAE, with abnormal vital signs, abnormal physical examination findings, abnormal oral examination findings, abnormal laboratory tests results and abnormal 12-lead ECG readings | From baseline to Month12
  AE, SAE, vital signs, physical examination, oral examination, laboratory examination (blood routine, urine routine/urine sediment, blood biochemistry, coagulation function), 12-lead ECG
ADA positive rate and ADA titer (if applicable) | Baseline and Month 1, Month3, Month6, Month12
  ADA positive rate and ADA titer (if applicable)
NAb positive rate (if applicable) | Baseline and Month 1, Month3, Month6, Month12
  NAb positive rate (if applicable)

CONTACTS AND LOCATIONS:
Locations (1):
- Mabwell (Shanghai) Bioscience Co., Ltd., Beijing, China

IPD SHARING:
Plan to Share IPD: No